CLINICAL TRIAL: NCT04331613
Title: Safety and Efficacy Study of Human Embryonic Stem Cells Derived M Cells (CAStem) for the Treatment of Severe COVID-19 Associated With or Without Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Safety and Efficacy of CAStem for Severe COVID-19 Associated With/Without ARDS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Beijing YouAn Hospital (Other)
Responsible Party: Principal Investigator, Qi Zhou, Director, Institute of Zoology, Chinese Academy of sciences, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChineseASZQ-006
Record Dates: First submitted 2020-02-06; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-01

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome; Virus; Pneumonia; Acute Lung Injury
Keywords: CAStem; Stem Cells; Cell Therapy; IMRCs
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Pneumonia, Viral; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAStem (Experimental): A dose-escalation with 3 cohorts with 3 patients/cohort who receive doses of 3, 5 or 10 million cells/kg. If there is no safety concerns for each cohort, the dose will be escalated from lower dose to next higher dose.
  Interventions: Biological: CAStem

INTERVENTIONS:
Biological: CAStem — CAStem will be administered intravenously.

SUMMARY:
A phase1/2, open label, dose escalation, safety and early efficacy study of CAStem for the treatment of severe COVID-19 associated with or without ARDS.

DETAILED DESCRIPTION:
CAStem is an injectable product composed of immunity- and matrix-regulatory cells (IMRCs), also named M cells, differentiated from clinical-grade human embryonic stem cells (hESCs) will be expanded, harvested, and formulated at a concentration of 50 x 10^6 cells/mL. CAStem will be cryopreserved and transported to clinical site using liquid nitrogen vapor shipping vessels (< -150ºC). Prior to injection, CAStem will be thawed to liquefy quickly, and then reconstituted in normal saline.In the present study, the intravenous infusion dose of CAStem will be 3, 5 or 10 million cells/kg.

ELIGIBILITY:
Inclusion criteria:

1. Chinese patients, aged 18 to 70 years old, males or females;
2. Diagnosis of COVID-19, and confirm by chest CT scan;
3. According to the diagnosis and treatment plan for the novel coronavirus disease (COVID-19) (trial version 5) issued by the National Health Commission (NHC) on the diagnostic criteria for severe or critical ill COVID-19 patients including the patients with acute respiratory distress syndrome (ARDS), the specific diagnostic criteria are:

   Severely ill patients should meet all of the following:
   * 1. Respiratory distress, RR ≥ 30 times/min.
   * 2. In a resting state (without oxygen supplementation), oxygen saturation ≤ 93%.
   * 3. Partial arterial oxygen pressure (PaO2) / oxygen absorption concentration (FiO2) ≤ 300 mmHg (1 mmHg = 0.133 kpa). High altitude (above sea level 1000 m) area should be calibrated for PaO2/FiO2 according to the following method: PaO2/FiO2*[atmospheric pressure (mmHg)/760]. Patients with obvious progress in lung lesions by chest CT within 24-48 hours should be counted as the server cases.

   Critically ill patients should meet one of the following :
   * 1. Respiratory failure, the mechanical ventilation required.
   * 2. Shock.
   * 3. Associated with other organ failure, ICU needed for monitoring and management.
4. Voluntarily participate in the study, agree to comply with the requirements of the clinical trial protocol, and sign the informed consent.

Exclusion criteria:

1. Patients with a history of transplantation of cells or organ(s).
2. Patients with a history of malignancy or pathology indicating severe atypical hyperplasia.
3. Patients without life expectancy of 48 hours.
4. Patients with moderate to severe liver failure (Childs Pugh scores > 12).
5. Patients with cardiogenic pulmonary edema.
6. Patients with a history of deep vein thrombosis or pulmonary embolism within 3 months before the screening.
7. Patients with severe chronic pulmonary diseases, including but not restricted to the patients with WHO grade III or IV pulmonary hypertension or those with chronic pulmonary diseases requiring long-term oxygen therapy.
8. Patients with unstable ventricular tachycardia or ventricular fibrillation.
9. Patients with poor coagulation, severe bleeding tendency or active bleeding at present.
10. Patients with serious dysfunction involved in the major organs or systems (liver, kidney, gastrointestinal, cardiovascular, blood coagulation, central system, etc.) besides the respiratory system are not suitable to participate in the present study.
11. Patients with a history of severe conditions in any organs or systems.
12. Patients who are unable to accept other invasive rescue except cardiopulmonary resuscitation.
13. Patients who are allergic to the main active ingredients or excipients of the investigational drug.
14. Women who are pregnant, breastfeeding or planning to become pregnant during the study period. Woman of childbearing age who is not willing to use appropriate contraceptive methods through the completion of the clinical study.
15. Patients whose participation is considered to bring significant risks to the present clinical study, cause confusion in analysis, or significantly interfere with the clinical research results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Adverse reaction (AE) and severe adverse reaction (SAE) | Within 28 days after treatment
  Frequency of adverse reaction (AE) and severe adverse reaction (SAE) within 28 days after treatment
Changes of lung imaging examinations | Within 28 days after treatment
  Evaluation by chest CT

SECONDARY OUTCOMES:
Time to SARS-CoV-2 RT-PCR negative | Within 28 days after treatment
  Marker for SARS-CoV-2
Duration of fever (Celsius) | Within 28 days after treatment
  The duration of a fever above 37.3 degrees Celsius
Changes of blood oxygen (%) | Within 28 days after treatment
  Marker for efficacy
Rate of all-cause mortality within 28 days | Within 28 days after treatment
  Marker for efficacy
Lymphocyte count (*10^9/L) | Within 28 days after treatment
  Counts of lymphocyte in a litre (L) of blood
Alanine aminotransferase (U/L) | Within 28 days after treatment
  Alanine aminotransferase in unit (U)/litre(L)
Creatinine (umol/L) | Within 28 days after treatment
  Creatinine in micromole (umol)/litre(L)
Creatine kinase (U/L) | Within 28 days after treatment
  Creatine kinase in U/L
C-reactive protein (mg/L) | Within 28 days after treatment
  C-reactive in microgram (mg)/litre(L)
Procalcitonin (ng/L) | Within 28 days after treatment
  Procalcitonin in nanogram (ng)/litre(L)
Lactate (mmol/L) | Within 28 days after treatment
  Lactate in millimole(mmol)/litre(L)
IL-1beta (pg/mL) | Within 28 days after treatment
  IL-1beta in picogram(pg)/millilitre(mL)
IL-2 (pg/mL) | Within 28 days after treatment
  IL-2 in pg/mL
IL-6 (pg/mL) | Within 28 days after treatment
  IL-6 in pg/mL
IL-8 (pg/mL) | Within 28 days after treatment
  IL-8 in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Qi, Doctor, Principal Investigator — Institute of Zoology, Chinese Academy of Sciences
Locations (1):
- Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing, China, China